CLINICAL TRIAL: NCT02858973
Title: A Phase 1B, Randomized, Placebo-Controlled, Double-Blind, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Q203 When Administered Orally to Healthy Adult Subjects
Brief Title: A Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of Multiple Doses of Q203 in Normal Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q203-TB-PI-US002
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — telacebec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q203 (Experimental): Q203 tablets
  Interventions: Drug: Q203
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q203
  Arms: Q203
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is randomized, double-blind, placebo-controlled, multiple ascending dose study of Q203 in healthy volunteers conducted at one study center in the United States

DETAILED DESCRIPTION:
Six (6) cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation. In each cohort, subjects will receive multiple oral doses of Q203 or placebo for 14 days QD with a standard meal. Subjects will participate in only one cohort.

Safety (i.e., physical examinations, vital signs, ECGs, clinical laboratory tests, and adverse events [AEs]) will be assessed throughout the study; serial blood and urine samples will be collected for these assessments. Blood samples will also be collected for the PK assessment of Q203.

Escalation to the next dose level (i.e., initiation of the next cohort) will not take place until the Principal Investigator (PI), medical monitor, and representatives of the Sponsor have reviewed all available safety and tolerability from the previous cohorts and agree to the initiation of the next cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.
2. Healthy adult male and/or female (non-childbearing potential only), 19 to 55 years of age, inclusive, at screening.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Safety assessment through adverse event, vital signs, ECG, laboratory results, and telemetry monitoring | 16 days post dose

SECONDARY OUTCOMES:
Pharmacokinetic analysis: Area under the curve | 16 days post dose
Pharmacokinetic analysis: Maximum observed plasma drug concentration | 16 days post dose
Pharmacokinetic analysis: Time of maximum observed concentration | 16 days post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No